CLINICAL TRIAL: NCT01950572
Title: Tissue Procurement and Natural History Study of Patients With Malignant Mesothelioma and Other Mesothelin Expressing Cancers
Brief Title: Tissue Procurement and Natural History Study of Patients With Malignant Mesothelioma
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130202; 13-C-0202
Record Dates: First submitted 2013-09-21; First posted 2013-09-25 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-12-17

CONDITIONS: Mesothelioma; Thymoma; Pancreatic Neoplasms; Biliary Tract Neoplasms; Stomach Neoplasms
Keywords: Samples; Biobank; Lung Neoplasms; Ovarian Neoplasms; Natural History
MeSH Terms: conditions — Mesothelioma; Thymoma; Pancreatic Neoplasms; Biliary Tract Neoplasms; Stomach Neoplasms; Lung Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Eligible cancer diagnosis: Subjects with mesothelioma, thymic carcinoma, pancreatic or biliary adenocarcinoma or lung, gastric or ovarian cancers

SUMMARY:
Background:

* Malignant mesothelioma is a malignancy arising from the mesothelial cells of the pleura, peritoneum, pericardium, or tunica vaginalis.
* Mesothelioma accounts for 0.10% of deaths annually in the United States. Malignant pleural mesothelioma is the most common of these, comprising of 80% of the cases with an annual incidence of about 2,500 in the United States.
* The median survival from diagnosis of pleural mesothelioma is approximately 12 months. The majority of patients present with stage III or IV disease with 85-90% of patients considered unresectable at diagnosis.
* Peritoneal mesothelioma has a better prognosis than pleural mesothelioma; nevertheless, patients undergoing therapy for peritoneal mesothelioma have few well-studied treatment options due in large part to the rarity of the disease.

Objectives:

-To allow sample acquisition for use in the study of mesothelioma.

Eligibility:

* All patients age greater than or equal to 2 years with malignant mesothelioma
* Must be able and willing to provide informed consent if 18 or over; parent or guardian must be able and willing to provide consent for patients under the age of 18

Design:

* Up to 1000 subjects will be enrolled.
* Patients will be followed to determine the course of disease and to record any treatment received for mesothelioma.
* Patients will undergo sampling of blood, urine, tumor and abnormal body fluids for tissue banking.
* Studies which may be performed on banked material include genetic and genomic studies, establishment of cell cultures and immunologic studies.

DETAILED DESCRIPTION:
Background:

* Malignant mesothelioma is a malignancy arising from the mesothelial cells of the pleura, peritoneum, pericardium, or tunica vaginalis.
* Mesothelioma accounts for 0.10% of deaths annually in the United States. Malignant pleural mesothelioma is the most common of these, comprising of 80% of the cases with an annual incidence of about 2,500 in the United States.
* The median survival from diagnosis of pleural mesothelioma is approximately 12 months. The majority of patients present with stage III or IV disease with 85-90% of patients considered unresectable at diagnosis.
* Peritoneal mesothelioma has a better prognosis than pleural mesothelioma; nevertheless, patients undergoing therapy for peritoneal mesothelioma have few well-studied treatment options due in large part to the rarity of the disease.
* In addition to mesothelioma, mesothelin is highly expressed in several cancers, including pancreatic, biliary adenocarcinomas, gastric and ovarian cancers; mesothelin is also expressed in a significantly larger proportion of thymic carcinoma than thymoma.
* Mesothelin expression level has been correlated with improved overall survival in thymic cancer and with reduced overall survival in patients with lung cancer.

Objective:

-To allow sample acquisition for use in the study of mesothelioma and other mesothelin expressing cancers.

Eligibility:

* All participants age greater than or equal to 2 years with malignant mesothelioma
* All participants age greater than or equal to 18 years with thymic carcinoma, pancreatic or biliary adenocarcinoma or lung, gastric or ovarian cancers
* Must be able and willing to provide informed consent if 18 or over; parent or guardian must be able and willing to provide consent for participants under the age of 18

Design:

* Up to 1000 participants will be enrolled.
* Participants will be followed to determine the course of disease and to record any treatment received for the eligible mesothelin expressing cancer.
* Participants will undergo sampling of blood, urine, tumor and abnormal body fluids for tissue banking.
* Studies which may be performed on banked material include genetic and genomic studies, establishment of cell cultures and immunologic studies.

ELIGIBILITY:
* INCLUSION CRITERIA:
* All participants greater than or equal to 2 years of age with malignant mesothelioma.
* All participants greater than or equal to18 years of age with thymic carcinoma, pancreatic or biliary adenocarcinoma or lung, gastric or ovarian cancers.
* Confirmed pathological diagnosis is required
* Ability and willingness of participant to provide informed consent to participation.

EXCLUSION CRITERIA:

* Active symptomatic major organ disorder that would increase the risk of biopsy, including but not limited to ischemic heart disease, recent myocardial infarction, active congestive heart failure, pulmonary dysfunction.
* Pregnant women
* Active concomitant medical or psychological illnesses that may increase the risk to the participant or in adult participants, inability to obtain informed consent, at the discretion of the principal investigator.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons with a diagnosis of any of the thoracic or GI cancers under study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-09-09 (Actual); Primary Completion 2033-07-25 (Estimated)

PRIMARY OUTCOMES:
sample aquisition | Ongoing
  allow sample acquisition for use in the study of mesothelioma

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data in BTRIS will be shared throughout the course of the study and indefinitely with the permission of the investigator.@@@@@@Genomic data will be shared from the time of upload to genomic database.
Access Criteria: Clinical IPD will be shared through the BTRIS database for open ended analysis. All BTRIS subscribers, generally limited to the NIH Clinical Center, may request data.@@@@@@Genomic IPD will be shared through dbGaP, per rules of the database, for purposes of genomic analysis.

REFERENCES:
- [Derived] Mian I, Abdullaev Z, Morrow B, Kaplan RN, Gao S, Miettinen M, Schrump DS, Zgonc V, Wei JS, Khan J, Pack S, Hassan R. Anaplastic Lymphoma Kinase Gene Rearrangement in Children and Young Adults With Mesothelioma. J Thorac Oncol. 2020 Mar;15(3):457-461. doi: 10.1016/j.jtho.2019.11.011. Epub 2019 Nov 26. PMID 31783178
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-C-0202.html